CLINICAL TRIAL: NCT00096174
Title: Phase II Study of C225 (Erbitux or Cetuximab) in Combination With Cisplatin and Definitive Radiation in Unresectable Stage IV Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase II Study of Concurrent C225, Cisplatin and Radiation in Stage IV Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000390923; U10CA021115 (NIH); E3303 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Platinum; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin, C225, Radiation (Experimental): * Cetuximab therapy: Patients receive an initial loading dose of cetuximab intravenously (IV) over 2 hours on day 1. Patients then receive cetuximab IV over 1 hour on days 8, 15, 22, 29, 36, 43, 50, and 57.
  * Chemoradiotherapy: Beginning on day 15 of cetuximab therapy, patients undergo radiotherapy once daily, 5 days a week, for at least 7 weeks. Patients also receive cisplatin IV over 1-2 hours on days 15, 36, and 57.
  * Cetuximab maintenance therapy: After the completion of chemoradiotherapy, patients continue to receive cetuximab IV over 1 hour once weekly for 6-12 months.
  Interventions: Biological: cetuximab C225; Drug: cisplatin; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab C225 — 400 mg/m^2 IV over 120 minutes on Day 1, 250 mg/m^2 IV over 60 minutes on Day 8, then weekly
  Other Names: Cetuximab; Erbitux
Drug: cisplatin — 75 mg/m^2 IV over 30-60 minutes starting day 15 every 3 weeks * 3 (Days 1, 22, and 43 of radiation therapy (RT))
  Other Names: Platinol; Platinol-AQ; CDDP; DDP; DACP; Platinum; cis-Platinum
Radiation: radiation therapy — RT 70 Gy / 35 starting Day 15, 200cGy / d * 7 weeks (35 fractions)

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Cetuximab may make the tumor cells more sensitive to radiation therapy and chemotherapy. Giving monoclonal antibody therapy together with chemoradiotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab and cisplatin together with radiation therapy works in treating patients with locally advanced or regional stage IV head and neck cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine 2-year progression-free survival in patients with unresectable locally advanced or regional stage IV squamous cell or undifferentiated carcinoma of the head and neck treated with cetuximab, cisplatin, and definitive radiotherapy.

Secondary

* Determine response rate and overall survival in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Correlate epidermal growth factor receptor (EGFR) expression by immunohistochemistry, EGFR phosphorylation, map kinase, Akt, signal transducer and activator of transcription 3 (STAT3), and other tissue and serum tests with toxicity of this regimen and outcomes in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor site (hypopharynx vs. oropharynx vs. oral cavity vs. larynx), primary tumor stage (T1-3 vs. T4), and nodal status (N0 vs. N1 vs. N2-3).

* Cetuximab therapy: Patients receive an initial loading dose of cetuximab IV over 2 hours on day 1. Patients then receive cetuximab IV over 1 hour on days 8, 15, 22, 29, 36, 43, 50, and 57.
* Chemoradiotherapy: Beginning on day 15 of cetuximab therapy, patients undergo radiotherapy once daily, 5 days a week, for at least 7 weeks. Patients also receive cisplatin IV over 1-2 hours on days 15, 36, and 57.
* Cetuximab maintenance therapy: After the completion of chemoradiotherapy, patients continue to receive cetuximab IV over 1 hour once weekly for 6-12 months.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 10 years.

ACCRUAL: A total of 69 patients were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell or undifferentiated carcinoma of the head and neck (excluding nasopharynx, paranasal sinus, and parotid gland)

  * Unresectable locally advanced or regional stage IV disease
  * No evidence of distant metastases
* Must have demonstrable primary tumor site
* Measurable disease
* Unresectable disease

  * Meets the following criteria for unresectable disease by tumor site:

    * Hypopharynx, meeting 1 of the following criteria:

      * Extension across the midline of the posterior pharyngeal wall
      * Any evidence of fixation to the cervical spine
    * Larynx

      * Direct subglottic extension (>3cm) into surrounding muscle or skin
    * Oral cavity

      * Lesion precluding functional reconstruction
    * Base of tongue, meeting 1 of the following criteria:

      * Extension into the root of the tongue
      * Patient refuses total glossectomy
    * Tonsillar area, meeting 1 of the following criteria:

      * Extension into pterygoid area as manifested by x-ray or trismus
      * Extension across midline of pharyngeal wall
      * Direct extension into soft tissue of the neck
    * Unilateral neck node metastases fixed to carotid artery, mastoid, base of skull, or cervical spine with any of the above tumors
* Patients requiring total glossectomy are eligible
* Age>=18 years
* ECOG Performance status of 0-1
* Adequate hematologic, renal, and hepatic function obtained <=4 weeks prior to registration

  * Absolute neutrophil count ≥ 2,000/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Hemoglobin ≥ 9.0 g/dL
  * Alkaline phosphatase ≤ 3 times normal
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 3 times normal
  * Bilirubin ≤ 1.5 mg/dL
  * Creatinine ≤ 1.2 mg/dL OR creatinine clearance ≥ 50 mL/min
* Able to tolerate fluid load
* At least 14 days since major surgery (including dental extraction) except percutaneous endoscopic gastrostomy (PEG) placement or mediport placement

Exclusion Criteria:

* Pregnant or nursing
* Fertile patients do not use effective contraception
* Patients who refuse surgery but whose tumors are technically resectable OR whose tumors are unresectable for medical reasons are not eligible
* Disease metastases below the clavicles or elsewhere (M1) or with a postoperative recurrence
* Prior excisional surgery of head and neck tumor
* Prior radiotherapy to the head and neck region
* Prior chemotherapy
* Prior drugs that target the epidermal growth factor receptor pathway
* Prior chimerized or murine monoclonal antibody
* Active systemic infection
* Known allergy to murine proteins
* Severe chronic obstructive pulmonary disease requiring ≥ 3 hospitalizations within the past year
* Myocardial infarction within the past 3 months
* Uncontrolled congestive heart failure
* Unstable or uncontrolled angina
* Clinically apparent jaundice
* Postoperative recurrence
* Other malignancy within the past 3 years except resected basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other in situ tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-04-08 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center

REFERENCES:
- [Result] Langer CJ, Lee JW, Patel UA, et al.: Preliminary analysis of ECOG 3303: concurrent radiation (RT), cisplatin (DDP) and cetuximab (C) in unresectable, locally advanced (LA) squamous cell carcinoma of the head and neck (SCCHN). [Abstract] J Clin Oncol 26 (Suppl 15): A-6006, 2008.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to accrual on 12/21/2004, accrued its first patient on April 8, 2005, and was closed on 07/20/2006. The final accrual was 69 patients.
Period: Overall Study
Arm/Group | Cisplatin, C225, Radiation
Started | 69
Began Protocol Therapy | 66 (3 patients never started treatment)
Eligible and Treated | 60 (6 treated patients were ineligible)
Completed | 7
Not Completed | 62
Not completed — Lack of Efficacy | 9
Not completed — Adverse Event | 15
Not completed — Death | 6
Not completed — Withdrawal by Subject | 15
Not completed — Not started protocol therapy | 3
Not completed — Ineligible | 6
Not completed — other reason | 8

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin, C225, Radiation
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 54.8 [42.0 to 78.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-free Survival Rate
Description: Two-year progression-free survival rate was defined as the proportion of patients that were alive progression-free two years after registration into the study. Disease progression was assessed per modified RECIST criteria, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, in either primary or nodal lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of new lesions. Kaplan-Meier estimate of 2-year progression-free survival was calculated in the 60 eligible and treated patients.
Time Frame: assessed every 3 months for 2 years
Population: Eligible and treated
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cisplatin, C225, Radiation
Number analyzed (Participants) | 60
proportion of participants | 47 [33 to 61]

2. Secondary Outcome: 2-year Overall Survival Rate
Description: Overall survival was defined as time from registration to death from any cause. Patients alive at last follow-up were censored. The 2-year overall survival rate was defined as the percentage of patients that were still alive two years after registration into the study. Kaplan-Meier estimate of 2-year overall survival was calculated in the 60 eligible and treated patients.
Time Frame: assessed very 3 months for 2 years
Population: Eligible and treated
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cisplatin, C225, Radiation
Number analyzed (Participants) | 60
proportion of participants | 66 [54 to 78]

3. Secondary Outcome: Overall Response Rate
Description: Response was assessed per Response Evaluation in Solid Tumor (RECIST) criteria by physical assessment and CT. Overall response = complete response (CR) + partial response (PR). CR was defined as the disappearance of all target and non-target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters of target lesions, along with non-progressive disease of non-target lesions. Overall response rate (i.e., proportion of patients who had CR or PR) and the corresponding 90% confidence intervals were calculated for the 60 eligible and treated patients
Time Frame: assessed after all chemoradiation therapy completed Week 9, then every 3 months on C225 maintenance therapy, and every 3 months for 2 years, every 6 months post-treatment 2 years from study entry
Population: Eligible and treated
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Cisplatin, C225, Radiation
Number analyzed (Participants) | 60
proportion of participants | 66.7 [55.3 to 76.7]

ADVERSE EVENTS:
Time Frame: Assessed weekly while on treatment, and every 3 months for 2 years
Arm/Group | Cisplatin, C225, Radiation
Serious Adverse Events (participants affected / at risk) | 64/66
Other Adverse Events (participants affected / at risk) | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin, C225, Radiation (N=66)
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 1
Hearing w/w-o audiogr not in monitor prg (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Leukopenia (Investigations) | 19
Lymphopenia (Investigations) | 2
Neutrophenia (Investigations) | 17
Thrombocytopenia (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 4
Fatigue (General disorders) | 15
Fever w/o neutropenia (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Weight loss (Investigations) | 18
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 17
Radiation dermatitis (Injury, poisoning and procedural complications) | 12
Wound - non-infectious (Injury, poisoning and procedural complications) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 23
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 13
Dental problems (Gastrointestinal disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 30
Esophagitis (Gastrointestinal disorders) | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 4
Muco/stomatitis by exam, pharynx (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) anus (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 36
Salivary problems (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 6
Larynx, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
ALT increased (Hepatobiliary disorders) | 1
AST increased (Hepatobiliary disorders) | 2
Bilirubin increased (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3
Creatinine increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 13
Hyponatremia (Metabolism and nutrition disorders) | 14
Trismus (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Neuropathy-motor (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Ocular-other (Eye disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Chest/thoracic pain NOS (Cardiac disorders) | 1
Esophagus, pain (Gastrointestinal disorders) | 1
Head/headache (Nervous system disorders) | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 2
Oral cavity, pain (Gastrointestinal disorders) | 5
Pain NOS (General disorders) | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 2
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1
Infection Gr0-2 neut, abdomen (Infections and infestations) | 1
Infection Gr0-2 neut, foreign body (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 2
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 3
Infection Gr0-2 neut, skin (Infections and infestations) | 4
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Infection w/ unk ANC bronchus (Infections and infestations) | 1
Infection w/ unk ANC conjunctiva (Infections and infestations) | 1
Infection w/ gr3-4 neut, blood (Infections and infestations) | 1
Infection Gr0-2 neut, blood (Infections and infestations) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin, C225, Radiation (N=66)
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 5
Anemia (Blood and lymphatic system disorders) | 60
Leukopenia (Investigations) | 55
Neutropenia (Investigations) | 34
Thrombocytopenia (Investigations) | 20
Hypotension (Vascular disorders) | 12
Fatigue (General disorders) | 55
Fever w/o neutropenia (General disorders) | 15
Insomnia (Psychiatric disorders) | 8
Rigor/chills (General disorders) | 4
Weight loss (Investigations) | 57
Burn (Injury, poisoning and procedural complications) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 29
Alopecia (Skin and subcutaneous tissue disorders) | 15
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7
Rash: ache/acneiform (Skin and subcutaneous tissue disorders) | 58
Radiation dermatitis (Injury, poisoning and procedural complications) | 18
Skin-other (Skin and subcutaneous tissue disorders) | 31
Anorexia (Gastrointestinal disorders) | 45
Constipation (Gastrointestinal disorders) | 33
Dehydration (Metabolism and nutrition disorders) | 12
Dental problems (Gastrointestinal disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 21
Dry mouth (Gastrointestinal disorders) | 38
Dysphagia (Gastrointestinal disorders) | 48
Dyspepsia (Gastrointestinal disorders) | 9
Muco/stomatitis by exam, oral activity (Gastrointestinal disorders) | 5
Muco/stomatitis (symptom) oral activity (Gastrointestinal disorders) | 59
Nausea (Gastrointestinal disorders) | 50
Salivary problems (Gastrointestinal disorders) | 26
Taste disturbance (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 34
Infection Gr0-2 neut,oral cavity (Infections and infestations) | 6
Infection Gr0-2 neut,skin (Infections and infestations) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 49
Alkaline phosphatase (Investigations) | 23
ALT increased (Hepatobiliary disorders) | 34
AST increased (Hepatobiliary disorders) | 26
Bilirubin (Hepatobiliary disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 24
Creatinine (Investigations) | 18
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 46
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 30
Hypernatremia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 47
Dizziness (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 11
Neutropathy-sensory (Nervous system disorders) | 8
Abdomen,pain (Gastrointestinal disorders) | 11
Head/headache (Nervous system disorders) | 13
Middle ear, pain (Ear and labyrinth disorders) | 6
Oral cavity, pain (Gastrointestinal disorders) | 18
Skin, pain (Skin and subcutaneous tissue disorders) | 4
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 5
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 4
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No